CLINICAL TRIAL: NCT02304627
Title: Effect of Food on the Pharmacokinetics of NNC0123-0000-0338 in a Tablet Formulation in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1953-3974; 2014-000979-87 (EudraCT Number); U1111-1154-0535 (Other: WHO)
Record Dates: First submitted 2014-11-21; First posted 2014-12-02 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Eating meal immediately after dosing (Experimental)
  Interventions: Drug: insulin 338 (GIPET I)
- Eating meal 30 min after dosing (Experimental)
  Interventions: Drug: insulin 338 (GIPET I)
- Eating meal 1 hour after dosing (Experimental)
  Interventions: Drug: insulin 338 (GIPET I)
- Eating meal 6 hour after dosing (Experimental)
  Interventions: Drug: insulin 338 (GIPET I)

INTERVENTIONS:
Drug: insulin 338 (GIPET I) — Each subject will be randomly allocated to a fixed treatment sequence of four single-dose administrations of oral insulin 338 in a GIPET® I tablet, administered on four separate dosing visits. The subjects will be dosed in the morning in the fasting state prior to four different post-dose fasting periods.

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the effect of food on the pharmacokinetics (the exposure of the trial drug in the body) of NNC0123-0000-0338 in a tablet formulation in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64 years (both inclusive) at the time of signing informed consent
* Body mass index 18.5-28.0 kg/m^2 (both inclusive)
* Subject who is considered to be healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products
* Previous participation in this trial. Participation is defined as informed consent
* Presence of clinically significant acute and chronic gastrointestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea) within 2 weeks prior to first dosing, as judged by the investigator

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-11-24 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin 338 concentration-time curve | From a 0-288 hours NNC0123-0000-0338 serum concentration-time-curve based on 41 sampling time points

SECONDARY OUTCOMES:
Area under the serum insulin 338 concentration-time curve | From 0 to 288 hours after a single dose (SD)
Maximum observed serum insulin 338 concentration | From 0 to 288 hours after a single dose (SD)
Area under the plasma capric acid concentration-time curve | From 0 to 24 hours after a single dose
Maximum observed plasma capric acid concentration | From 0 to 24 hours after a single dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Halberg IB, Lyby K, Wassermann K, Heise T, Plum-Morschel L, Zijlstra E. The Effect of Food Intake on the Pharmacokinetics of Oral Basal Insulin: A Randomised Crossover Trial in Healthy Male Subjects. Clin Pharmacokinet. 2019 Nov;58(11):1497-1504. doi: 10.1007/s40262-019-00772-2. PMID 31093929
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com